CLINICAL TRIAL: NCT02493101
Title: Potential of Periostin as a Tissue and Urinary Biomarker in Lupus Nephritis and IgA Nephropathy Patients
Brief Title: The Correlation of Periostin and Renal Pathology in Chronic Kidney Disease Patients
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Collaborators: Thailand Research Fund (Other)
Responsible Party: Sponsor
Other Study IDs: IRBRTA1168/2556
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Lupus Nephritis; IgA Nephropathy
Keywords: Periostin staining; Urine periostin level; Lupus nephritis; IgA nephropathy
MeSH Terms: conditions — Lupus Nephritis; Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — urine and kidney tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Chronic kidney disease: Patients with lupus nephritis and IgA nephropathy
- Control: Healthy controls

SUMMARY:
The purpose of this study is to determine the location of periostin and urine periostin level in patients with lupus nephritis and IgA nephropathy.

DETAILED DESCRIPTION:
Total of 50 lupus nephritis and IgA nephropathy patients who met the inclusion criteria were included in this study. The information sheet and informed consent will be obtained before collecting the patient's data. All patients were interviewed for collecting demographic data and laboratory testing were reviewed from patient's record. Kidney tissue and urine sample were collected at the biopsy date from patients.Kidney tissue were stained with hematoxylin and eosin (H&E), Masson's trichrome solution and immunohistochemistry for periostin. The location of periostin staining in kidney tissue were assessed by renal pathologist.

The total of 50 urine samples from patients and 50 urine samples from healthy controls were measured for periostin level by enzyme-linked immunosorbent assay. The Mann-Whitney rank-sum test was used for comparing urine periostin level between patients and healthy controls and also other variables between patients with urine periostin detection and without urine periostin detection. Spearman correlation coefficients were used test correlations between urine periostin level in patients and other variables. Receiver operating characteristic curves was generated to calculate the area under the curve and find the best cutoff value of urine periostin level for distinguishing patients from healthy controls. P-values < 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years
* at least three glomeruli obtained at biopsy

Exclusion Criteria:

* Patients with urinary tract obstruction
* Patients with urinary tract infection
* Patients with kidney transplant
* Patients with cancer diseases
* Patients with asthma
* Patients with advanced heart disease
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting at the Department of Medicine, Phramongkutklao Hospital, Bangkok, Thailand
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Urine periostin level in lupus nephritis and IgA nephropathy patients compared with healthy controls | 2 years

SECONDARY OUTCOMES:
Correlation of urine periostin level in lupus nephritis and IgA nephropathy patients and other variables | 2 years
The best cutoff value of urine periostin level for distinguishing patients from healthy controls | 2 years
The variables that involved in urine periostin detection in lupus nephritis and IgA nephropathy patients | 2 years
Periostin staining in kidney tissue from lupus nephritis and IgA nephropathy patients | 2 years